CLINICAL TRIAL: NCT03630185
Title: A Prospective Randomized-controlled Trial of Custom-manufactured vs. Off-the-rack (OTR) Compression Hosiery for Initial Management of Venous Disease
Brief Title: A Comparison of Custom-manufactured vs. Off-the-rack (OTR) Compression Hosiery for Initial Management of Venous Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not reach the enrollment goal.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Stuart A Harlin, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-17-0015
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Venous Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Custom-manufactured compression hosiery (Isobar) (Experimental): The custom-fitted garment is manufactured specifically for each patient based on measurements taken with a 3-dimensional volumetric laser scan of the extremity, and can be sized individually to each limb.
  Interventions: Device: Custom-manufactured compression hosiery (Isobar)
- Off-the-rack stockings (Sigvaris) (Active Comparator): Currently available off-the-rack compression hosiery are manufactured in eight fixed sizes (S-XLFC) that cannot be varied in size over their length to accommodate unusual anatomic patterns (eg., small ankle with large calf or vice versa) and may not achieve a comfortable fit that meets the compression goal over a uniform distribution of the limb.
  Interventions: Device: Off-the-rack stockings (Sigvaris)

INTERVENTIONS:
Device: Custom-manufactured compression hosiery (Isobar) — The custom-fitted garment is manufactured specifically for each patient based on measurements taken with a 3-dimensional volumetric laser scan of the extremity, and can be sized individually to each limb.
  Arms: Custom-manufactured compression hosiery (Isobar)
Device: Off-the-rack stockings (Sigvaris) — Currently available off-the-rack compression hosiery are manufactured in eight fixed sizes (S-XLFC) that cannot be varied in size over their length to accommodate unusual anatomic patterns (eg., small ankle with large calf or vice versa) and may not achieve a comfortable fit that meets the compression goal over a uniform distribution of the limb.
  Arms: Off-the-rack stockings (Sigvaris)

SUMMARY:
The purpose of this research study is to assess the efficacy of custom-manufactured compression hosiery (also known as compression stockings) compared to similar off-the-rack (OTR) compression stockings.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and sign an informed consent and complete study questionnaires
* Patient is participating in usual work and home activities with no changes anticipated for the duration of the study
* The use of compression stocking is prescribed in accordance with the usual practice and management of venous disorders
* The patient will confirm they are willing to pay for the compression stockings.

Exclusion Criteria:

* The patient has a known allergy to any component of the stocking (latex, etc)
* The patient has non-venous source of pain in either leg that could, in the opinion of the investigator, confound the results of the study i.e.Neuropathy, Arterial insufficiency, Diabetes
* The patient is confined to bed
* The patient has uncontrolled Congestive Heart Failure
* The patient has acute dermatitis
* The patient has weeping dermatosis
* Patients with venous ulcers will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Harlin, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Started | 4 | 4
30 Day Follow up | 1 | 1
90 Day Follow up | 0 | 1
6 Month Follow up | 0 | 0
Completed | 0 | 0
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar) | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (4.2) | 58.5 (12.5) | 63.75 (8.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 0 | 4 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1 | 0 | 1
  Hispanic | 1 | 0 | 1
  White | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pain Management Experienced During Their Postoperative Care as Assessed by Five-point Satisfaction Scale
Description: Five-point satisfaction scale consists of patients rating their overall postoperative pain management experience using a 5-point rating system. The scale ranges from 1 to 5, with 1 being "extremely dissatisfied", 2 "somewhat dissatisfied", 3 "Neutral/Neither satisfied nor dissatisfied", 4 "somewhat satisfied" and 5 "extremely satisfied" with their postoperative pain care.
Time Frame: 6 weeks
Population: Data was not collected for this outcome measure.
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Pain Management Experienced During Their Postoperative Care as Assessed by Five-point Satisfaction Scale
Description: as for outcome 1
Time Frame: 90 days
Population: Data was not collected for this outcome measure.
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Pain Management Experienced During Their Postoperative Care as Assessed by Five-point Satisfaction Scale
Description: as for outcome 1
Time Frame: 6 months
Population: Data was not collected for this outcome measure.
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Pain as Assessed by Brief Pain Inventory
Description: The Brief Pain Inventory is a medical questionnaire used to measure pain, developed by the Pain Research Group of the World Health Organization Collaborating Center for Symptom Evaluation in Cancer Care.
  The score is an average of seven questions about pain interference in life. The score scale is from 0 to 10. 0 being pain does not interfere and 10 being that it completely interferes. 10 would be a worst outcome.
Time Frame: Baseline
Population: Data was not collected for this outcome measure.
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Pain as Assessed by Brief Pain Inventory
Description: as for outcome 4
Time Frame: 6 weeks
Population: Data was not collected for this outcome measure.
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Pain as Assessed by Brief Pain Inventory
Description: as for outcome 4
Time Frame: 90 days
Population: Data was not collected for this outcome measure.
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Pain as Assessed by Brief Pain Inventory
Description: as for outcome 4
Time Frame: 6 months
Population: Data was not collected for this outcome measure.
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Overall Estimate of Functioning as Assessed by the SF-12 HRQoL Instrument (Overall HRQoL Estimate)
Description: The short-form 12 item (SF-12) HRQoL health status instrument measures Health-Related Quality of Life (HRQoL). It produces overall HRQoL estimates as well as sub-scale scores (Physical Component Summary (PCS) and Mental Component Summary (MCS)) that assess both mental/emotional and physical functioning related to health.
  The scoring scale is from 0 to 100, the higher the score the better the health related quality of life.
Time Frame: Baseline
Population: This data was not collected for 2 in the Off-the-rack stockings (Sigvaris) arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 2 | 4
score on a scale | 35.8 (10.0) | 45.8 (6.8)

9. Primary Outcome: Overall Estimate of Functioning as Assessed by the SF-12 HRQoL Instrument (Overall HRQoL Estimate)
Description: as for outcome 8
Time Frame: 30 days
Population: This data was not collected for 3 in the Off-the-rack stockings (Sigvaris) arm and 3 in the Custom-manufactured compression hosiery (Isobar) arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 1 | 1
score on a scale | 48.3 (0) | 44.0 (0)

10. Primary Outcome: Overall Estimate of Functioning as Assessed by the SF-12 HRQoL Instrument (Overall HRQoL Estimate)
Description: as for outcome 8
Time Frame: 90 days
Population: This data was not collected for 4 in the Off-the-rack stockings (Sigvaris) arm and 3 in the Custom-manufactured compression hosiery (Isobar) arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 1
score on a scale |  | 47.6 (0)

11. Primary Outcome: Overall Estimate of Functioning as Assessed by the SF-12 HRQoL Instrument (Overall HRQoL Estimate)
Description: as for outcome 8
Time Frame: 6 months
Population: This data was not collected for any in the Off-the-rack stockings (Sigvaris) arm or any in the Custom-manufactured compression hosiery (Isobar) arm.
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Physical Functioning as Assessed by the SF-12 HRQoL Instrument Physical Component Summary (PCS)
Description: as for outcome 8
Time Frame: Baseline
Population: This data was not collected for 2 in the Off-the-rack stockings (Sigvaris) arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 2 | 4
score on a scale | 32.5 (9.5) | 36.8 (3.7)

13. Primary Outcome: Physical Functioning as Assessed by the SF-12 HRQoL Instrument Physical Component Summary (PCS)
Description: as for outcome 8
Time Frame: 30 days
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 1 | 1
score on a scale | 29.9 (0) | 39.9 (0)

14. Primary Outcome: Physical Functioning as Assessed by the SF-12 HRQoL Instrument Physical Component Summary (PCS)
Description: as for outcome 8
Time Frame: 90 days
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 1
score on a scale |  | 36.3 (0)

15. Primary Outcome: Physical Functioning as Assessed by the SF-12 HRQoL Instrument Physical Component Summary (PCS)
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 11
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: Mental/Emotional Functioning as Assessed by the SF-12 HRQoL Instrument Mental Component Summary (MCS)
Description: as for outcome 8
Time Frame: Baseline
Population: This data was not collected for 2 in the Off-the-rack stockings (Sigvaris) arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 2 | 4
score on a scale | 39.2 (10.5) | 54.8 (10.7)

17. Primary Outcome: Mental/Emotional Functioning as Assessed by the SF-12 HRQoL Instrument Mental Component Summary (MCS)
Description: as for outcome 8
Time Frame: 30 days
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 1 | 1
score on a scale | 66.7 (0) | 48.1 (0)

18. Primary Outcome: Mental/Emotional Functioning as Assessed by the SF-12 HRQoL Instrument Mental Component Summary (MCS)
Description: as for outcome 8
Time Frame: 90 days
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 1
score on a scale |  | 58.8 (0)

19. Primary Outcome: Mental/Emotional Functioning as Assessed by the SF-12 HRQoL Instrument Mental Component Summary (MCS)
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 11
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Number of Patients Who Will be Progressing to Ablation Therapy
Description: Progression to ablation therapy will be determined by patient preference for further intervention.
Time Frame: 6 months
Population: Data was not collected for this outcome measure.
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Off-the-rack Stockings (Sigvaris) | Custom-manufactured Compression Hosiery (Isobar)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
Small sample size, did not reach target enrollment number.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT03630185/Prot_SAP_000.pdf